CLINICAL TRIAL: NCT04485624
Title: Do Children and Young People Attending the Paediatric Emergency Department Have Lower Levels of Vaccination Coverage Than Their Peers in the Local General Population?
Brief Title: Vaccination Coverage Amongst Children/Young People Attending the PED
Status: Completed | Type: Observational
Sponsor: Lancaster University (Other)
Collaborators: Pennine Acute Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Rachel Isba, Professor of Medicine and Consultant in Paediatric Public Health Medicine, Lancaster University
Other Study IDs: IRAS278815
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Vaccination/Immunisation Status
Keywords: Vaccination; Immunisation; Opportunistic; Child; Young person; Paediatric Emergency Department

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Attendees at Paediatric Emergency Department 1 (PED1): These participants will be recruited from the children and young people (under the age of 16) attending the PED of a large district general hospital.
  There was going to be a second group recruited but COVID meant that the site was not able to support non-COVID studies by the time the necessary approvals were in place.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
In the United Kingdom (UK), most childhood vaccinations are given in the community, although uptake has decreased in recent years. A Paediatric Emergency Department (PED) attendance offers an opportunity to check the vaccination status of children and young people (CYP) and all parents/carers should be asked about this routinely. Those not up-to-date with vaccinations could then be signposted to existing services or perhaps offered a vaccine in the PED.

CYP attending the PED may also have lower vaccination coverage than their peers, so may benefit even more from interventions to increase uptake. However, recall by parents/carers is not always sufficiently accurate to identify those who have not yet received all their age-appropriate vaccinations. The most complete record of an individual's vaccination history is held within their primary care records. However, these records are often in a separate computer system that is inaccessible from the hospital's main computer system, although some information (including vaccination) may be accessed from within the hospital via a third system.

This study aims to see if CYP attending the PED are under-vaccinated compared to their peers and assess the accuracy of parent/carer recall. The results of this study will then be used to inform recommendations for developing better ways to access accurate vaccination data during a PED consultation. If such a system existed, under-vaccinated children could be identified routinely during an attendance, and an intervention offered if appropriate. This would be particularly useful if there was an outbreak of a vaccine-preventable disease such measles.

All CYP (< 16 years old) attending a PED in a district general hospital in Manchester will be invited to participate. CYP/their parent/carer will be asked to provide consent for their vaccination records to be accessed as well as being asked if the child/young person is up-to-date with all their vaccinations. Approximately 1000 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* attending the study site PED; under the age of 16 at the time of attendance; able to give consent or accompanied by someone able to give consent

Exclusion Criteria:

* life threatening illness or injury

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and young people accessing PED
Sampling Method: Non-Probability Sample
Enrollment: 2693 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of children/young people attending the PED who have received all of their age-appropriate vaccinations. | Through study completion (estimated one year)
  The % of children and young people attending the PED who have received all of their age-appropriate vaccinations will be compared to their peers in the local general population.

SECONDARY OUTCOMES:
Accuracy of parent/carer recall of the vaccination status of children/young people attending the PED. | Through study completion (estimated one year)
  The accuracy of parent/carer recall of the vaccination status of children/young people attending the PED will be made by comparing their responses to electronic community records.
Percentage of children attending the PED who have received two doses of MMR by the age of 5 years. | Through study completion (estimated one year)
  The % of children attending the PED who have received two doses of the Measles, Mumps, and Rubella vaccine (MMR) by the age of 5 years will be compared to their peers in the local general population.
Percentage of children attending the PED who have received at least one dose of MMR by the age of 2 years. | Through study completion (estimated one year)
  The % of children attending the PED who have received at least one dose of MMR by the age of 2 years will be compared to their peers in the local general population.

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric Emergency Department, North Manchester General Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Results of study intended to be published in an open access journal within a year of completion of analysis of data.
  Anonymised data will be shared under certain circumstances; no patient-identifiable data will be available to other researchers.
Access Criteria: Anonymised data will be made available following reasonable request.

REFERENCES:
- [Derived] Isba R, Brennan L, Egboko F, Edge R, Davies N, Knight J. Unmet vaccination need among children under the age of five attending the paediatric emergency department: a cross-sectional study in a large UK district general hospital. BMJ Open. 2023 Jun 26;13(6):e072053. doi: 10.1136/bmjopen-2023-072053. PMID 37369415